CLINICAL TRIAL: NCT05402332
Title: A Phase 2b, Multicenter, Randomized, Double-blind, Placebo-Controlled, Crossover, Trial Assessing the Efficacy, Safety, and Tolerability of AVTX-801 in Subjects With Phosphoglucomutase 1 Deficiency Related Congenital Disorders of Glycosylation (PGM1-CDG)
Brief Title: Evaluating the Efficacy and Safety of D-galactose in PGM1-CDG (AVTX-801)
Acronym: AVTX-801
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eva Morava-Kozicz (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor-Investigator, Eva Morava-Kozicz, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY-24-00424; 20-009499 (Other: CHOP); FCDGC 8402 (Other: Rare Diseases Clinical Research Network (RDCRN)); AVTX-801-PGM1-201 (Other: other)
Record Dates: First submitted 2022-05-28; First posted 2022-06-02 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: PGM1-CDG - Phosphoglucomutase 1-Related Congenital Disorder of Glycosylation
MeSH Terms: conditions — Glycogen Storage Disease XIV | interventions — Galactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AVTX-801, then Placebo (Experimental): Participants receive AVTX-801 1.5g/kg/day (in applesauce) during Treatment Period 1 and then placebo (in applesauce) during Treatment Period 2.
  Interventions: Drug: AVTX-801; Drug: Placebo
- Placebo, then AVTX-801 (Experimental): Participants receive placebo (in applesauce) during Treatment Period 1 and then AVTX-801 1.5g/kg/day (in applesauce) during Treatment Period 2.
  Interventions: Drug: AVTX-801; Drug: Placebo

INTERVENTIONS:
Drug: AVTX-801 — D-Galactose medical grade supplement - 1.5g/kg/day (not to exceed 50 g/day)
  Other Names: D-Galactose
Drug: Placebo — placebo equivalent

SUMMARY:
This is a clinical trial to evaluate the efficacy of AVTX-801 (D-galactose) on the clinical manifestations of PGM1-CDG in participants currently taking D-galactose.

DETAILED DESCRIPTION:
Participants who sign consent will be screened for enrollment, and if they meet all eligibility criteria, they will enter a 4-week Run-In period. During the Run-In period, participants will continue to take D-galactose therapy, and will be monitored for hypoglycemic events, to establish a baseline rate. Following completion of the Run-In period participants will complete Baseline Day 1 procedures for treatment period 1 and be randomized in a 1:1 fashion to one of two treatment sequences: 1) AVTX-801 (plus applesauce) 1.5 g/kg/day (not to exceed 50 g/day) (treatment period 1) followed by placebo (plus applesauce ) (treatment period 2) or 2) Placebo (plus applesauce) (treatment period 1) followed by AVTX-801 (plus applesauce) 1.5 g/kg/day (not to exceed 50 g/day) (treatment period 2).

Each treatment period will end upon completion of 18 weeks of treatment or upon occurrence of a PGM1-CDG related event. There will be an open label recovery period of 18 weeks separating the two treatment periods, during which time the subject will receive commercially available D-galactose.

During the double-blind period of the study, participants will be closely monitored for clinical signs and symptoms related to or suspected to be related to withdrawal of D galactose therapy; specifically, recurrent or prolonged hypoglycemia, elevation of ALT and decreases in ATIII.

Upon completion of the double-blind portion of the study (i.e., either completion of both 18-week double-blind periods or occurrence of a PGM1-CDG related event during treatment period 2), participants will be permitted to enter a long-term, open-label, safety follow-up period of 12 months with AVTX-801.

ELIGIBILITY:
Inclusion Criteria

1. Subject is aged 18 to 60 years.
2. Subject has biologically and genetically proven PGM1-CDG.
3. Subject is currently on a stable dose of D-galactose therapy.
4. Non-pregnant, non-lactating female subjects of childbearing potential who are heterosexually active and non-sterile male subjects with female sexual partners of childbearing potential agree to use a highly effective method of contraception for the duration of the study, including the long-term safety follow-up period. A highly effective method of birth control is defined as one that results in a low failure rate (i.e., <1% per year) when used consistently and correctly, such as oral/injectable/inserted/implanted/transdermal contraceptives, condom with diaphragm, condom with spermicide, diaphragm with spermicide, intrauterine hormone- releasing system, or intrauterine device (IUD), or sexual abstinence. Contraception is not required where at least 6 weeks have passed since sterilization, defined as females having undergone one of the following surgeries: hysterectomy, bilateral tubal ligation or occlusion, bilateral oophorectomy, or bilateral salpingectomy; and males who are vasectomized. Contraception is not required where females are postmenopausal (defined as 12 consecutive months of spontaneous amenorrhea and age ≥51 years).
5. Subject/legally authorized representative (LAR) is able to understand and provide written informed consent, and assent (as applicable) to participate in this study.

Exclusion Criteria

1. Subject has aldolase B deficiency, galactosemia, hemolytic uremic syndrome, or severe anemia.
2. In the site Principal Investigator's opinion, subject has a history of galactose intolerance that precludes the subject from participation in this study.
3. In the site Principal Investigator's opinion, subject has previously experienced any of the following severe AEs from oral galactose:

   1. Severe diarrhea
   2. Severe, recurrent vomiting
   3. Constipation
   4. Galactosuria
   5. Increased liver glycogen storage.
4. Subject has any of the following:

   1. Liver failure
   2. ALT level >8x ULN
   3. AST level >8x ULN
5. Use of investigational compounds within the previous 6 months or current enrollment in another trial involving investigational compounds.
6. Subject is pregnant.
7. Subject has hepatic impairment that would require a dose adjustment, defined by the site Principal Investigator.
8. In the site Principal Investigator's opinion, subject is not able or willing to comply with the trial requirements.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2028-03-02 (Estimated); Study Completion 2028-03-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with at least one PGM1-CDG related event | after each treatment period (treatment periods are 18 weeks)
  Proportion of participants in each treatment group who experience at least one PGM1-CDG related event (recurrent or prolonged hypoglycemia, elevation of ALT and/or decrease in ATIII) during each treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Morava-Kozicz, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No